CLINICAL TRIAL: NCT06251570
Title: Evaluation of Dual Task Performance and Respiratory Muscle Endurance in Patients With Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslınur ÇAKIR, Physiotherapist, Hacettepe University
Other Study IDs: GO 23/56
Record Dates: First submitted 2024-01-04; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: Dual-task; lung cancer; respiratory muscle endurance
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Lung Cancer: Patients with Lung Cancer
  Interventions: Other: Evaluation of Dual Task Performance
- Control Group: Control Group
  Interventions: Other: Evaluation of Dual Task Performance

INTERVENTIONS:
Other: Evaluation of Dual Task Performance — The Montreal Cognitive Evaluation Scale will be used to evaluate the cognitive functions of the participants.
  Evaluation of Physical Activity Level: The Turkish validity and reliability of the International Physical Activity Questionnaire Short Form made by Sağlam et al. will be used.
  Evaluation of Quality of Life: It will be evaluated by the European Organization for Cancer Research and Treatments QLQ-C30 questionnaire.
  Fatigue Evaluation: A fatigue severity scale consisting of 9 items will be used.
  Dyspnea Assessment: The Modified Medical Research Council Dyspnea Scale will be used.
  Respiratory Muscle Endurance: Evaluation will be done by respiratory muscle endurance test at constant threshold load with a Power Breathe device and according to the metronome warning and a MOXY monitor will be used. In evaluation of dual-task performance, an auditory task test will be performed while walking on the treadmill.
  Other Names: Evaluation of Respiratory Muscle Endurance; Evaluation of Cognitive Function; Evaluation of Physical Activity Level; Evaluation of Quality of Life; Fatigue Evaluation; Dyspnea Assesment

SUMMARY:
Lung cancer is one of the most diagnosed cancer types worldwide, according to GLOBOCAN data published in 2020. According to these data, lung cancer comes second after breast cancer with 2,206,771 new diagnoses worldwide in 2020.

According to Türkiye's data for 2020, 41,264 new lung cancer diagnoses made. Lung cancer tumors are divide into two main histological groups non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC).

Current medical treatment methods for lung cancer are surgical resection, chemotherapy, radiotherapy, and targeted therapies. Cancer treatments can be administered as a combination of these methods appropriately selected for patients.

Advances in treatment methods in recent years have increased survival and prolonged life expectancy. However, these treatment methods may affect patients in various areas from functional independence to quality of life.

Cancer treatments can cause various cognitive impairments such as memory, executive functions, and concentration.

In particular, a significant number of cancer patients receiving chemotherapy report cognitive disturbances that include attention problems, memory loss, and mixed thought processes ('chemobrain' or 'chemofog?), often accompanied by mood disorders and fatigue.

Despite recent large cohort studies using neuropsychological testing and neuroimaging in cancer patients undergoing chemotherapy, it remains unclear whether cognitive deficits are due to treatment, cancer itself, and/or psychological factors.

Patients with cognitive impairment due to chemotherapy reported that they had difficulty performing and completing simple tasks such as preparing meals, keeping track of bills and paying, or getting ready to go out, and needed additional time to perform these tasks.

They may also find it difficult to perform necessary work-related tasks and then need to change jobs or cease employment altogether.

Therefore, treatment-related cognitive impairment can have a significant impact on cognitive, occupational, and social functioning, all of which can result in significant personal problems and, in many cases, reduced quality of life.

During daily activities, we often need to perform multiple tasks at the same time. These tasks are usually cognitive and motor tasks.

A dual-task is the simultaneous execution of two tasks that have different objectives and can performed independently. In this case, attention should be focused on two tasks at the same time. These tasks can be measured separately.

Deteriorated cognitive function due to cancer and its treatments can affect the dual-task performance of individuals in their daily lives and reduce their quality of life.

Respiratory symptoms can be seen in lung cancer and post-cancer survival. Cancer itself and treatments can affect the cardiorespiratory system.

Considering that the number of individuals living with lung cancer increases every year, the evaluation of dual-task performance and respiratory muscle endurance, which is related to the cognitive status of individuals, and if necessary, adding them to the rehabilitation program can reduce the symptoms of individuals and increase their quality of life.

DETAILED DESCRIPTION:
The aim of this study is to evaluate dual-task performance and respiratory muscle endurance in patients with lung cancer and compare them with healthy individuals.

H0: Dual-task performance and respiratory muscle endurance of patients with lung cancer are not different from healthy controls.

H1: Dual-task performance and respiratory muscle endurance values of patients with lung cancer are different from healthy controls.

Place and time of research:

Hacettepe University Faculty of Physical Therapy and Rehabilitation Cardiopulmonary It will be held in the Rehabilitation Unit. Between January 2024 and July 2024 It is planned to collect data and write the study.

Working Design:

Respiration as an outcome measure to determine the sample size of our study. Analysis was done according to muscle endurance. Analysis G*Power analysis system (G*Power Software version 3.1.9.3, Heinrich Heine University, Düsseldorf Germany) was made using For the power of our study to be 80%, at least 25 individuals with lung cancer should be included. 20% patient loss At least 30 lung cancer patients were included in the study, as was thought that will be. Age and gender-matched with the patient group, undiagnosed, 30 individuals consisting of volunteers will form the control group.

Individuals who will participate in the study are informed about the study verbally and in writing, An informed consent form will be obtained.

Research method and data collection tools:

Due to the COVID-19 pandemic, mask, distance, and hygiene rules will be followed to prevent transmission to or from participants. The patients will be taken into the study one by one and the measuring devices used after each patient will be disinfected and the unit will be ventilated.

All necessary infection control rules will be followed.

1. Demographic information: Participants' age, diagnosis, medical history, radiotherapy (number of days), chemotherapy (number of cures), occupation, body weight, height, BMI, history, family history, lifestyle characteristics (smoking, alcohol use), breathing stenosis, cough and sputum will be recorded.
2. Evaluation of Cognitive Function: The Montreal Cognitive Evaluation Scale (MOCA) will be used to evaluate the cognitive functions of the participants.

   MOCA was developed to measure different stages of cognitive impairment. It evaluates cognitive behaviors such as attention and concentration, executive functions, language, memory, visuospatial skills, abstract thinking and calculation. As memory tasks, recall from short-term memory, learning five words and recalling after five minutes; clock drawing test and three-dimensional cube painting as tasks requiring visuospatial skills; as tasks related to executive functions, tracing test, combining sequential number and letter patterns, verbal fluency and two-item abstract thinking task; sequential subtraction and forward-backward number space as attention, concentration, and working memory tasks; As language-related tasks, it includes questions about naming three pictures of animals, repeating two complex sentences, and time and place orientation.

   The highest possible score is 30 and the lowest score is 0. If the score is 21 and above, the cognitive level of the individual is considered normal.
3. Evaluation of Physical Activity Level: The Turkish validity and reliability of the International Physical Activity Questionnaire Short Form made by Sağlam et al. will be used.

   This questionnaire provides information on time spent in walking, moderate and vigorous physical activity. Time spent sitting is not included in the total score and is considered a separate question.

   The sum of moderate-intensity activity, vigorous activity, frequency of walking (days) and duration (minutes) is used to calculate the total score. The score in MET x minute units is obtained by multiplying the minute of activity with the MET score.

   For analysis of IPAQ data, it is calculated on walking: 3.3 METs, moderate-intensity physical activity: 4.0 METs, vigorous physical activity: 8.0 METs.

   People can be grouped according to their physical activity levels as 'inactive', 'minimally active', 'very active'.
4. Evaluation of Quality of Life: It will be evaluated by the European Organization for Cancer Research and Treatments (EORTC) QLQ-C30 questionnaire. The scale consists of the sub-headings of functional difficulties, general health status and symptom control and includes 30 questions.

   The lowest possible score is 0, and the highest score is 100. Its Turkish validity and reliability were evaluated by Cankurtaran friends in 2008.
5. Fatigue Evaluation: A fatigue severity scale consisting of 9 items will be used. The individual should answer the questions by thinking about the last week. Each item is scored between 1 and 7 in itself. 1 point indicates strongly disagree, 7 points strongly agree. The total score that can be obtained is a minimum of 9 and a maximum of 63. The scale score is the arithmetic mean of the total score obtained from nine items. As the scale score increases, the severity of fatigue increases. A total score of 36 and above or a scale score of 4 and above indicates severe fatigue in patients.
6. Dyspnea Assessment: The Modified Medical Research Council (MMRC) Dyspnea Scale will be used. The individual is asked to choose one of the 5 statements that best describe shortness of breath. A score of 0 indicates no shortness of breath except during vigorous exercise, while 4 points indicate that there is shortness of breath when getting out or getting dressed or undressing.
7. Evaluation of Respiratory Muscle Endurance: A Power Breathe device will be used in the evaluation of respiratory muscle endurance. Evaluation will be done by respiratory muscle endurance test at constant threshold load.

   The device we set with the value corresponding to 60% of the maximal inspiratory pressure will be placed in the mouth and the nose will be closed with a clip. The individual will be asked to breathe normally within the device for 10 minutes according to the metronome warning.

   Before applying the test, if the person feels too short of breath during the test, they will be informed that they can remove the device and thus the test will end. The result values will be obtained by multiplying the test time, the test time and the pressure value corresponding to the time.

   A MOXY monitor will be used to measure tissue oxygenation of the intercostal muscles during the test.
8. Evaluation of Dual-Task Performance: In evaluation of dual-task performance, an auditory task test will be performed while walking on the treadmill.

Patients will be asked to make choices on the computer based on the commands coming from the headphones while first standing on the treadmill, then walking at their preferred speed, and finally at speed higher than their preferred speed.

First, the speed preferred by individuals will be found. A progressive speed test will be used for this, in which the speed increases in 15 seconds. In order not to be affected by the numerical value, the speed part of the treadmill will be closed with the help of paper and hidden from the individual.

The participant will be asked to indicate when he has reached his preferred speed in each test. The average preferred walking speed will be found by averaging the preferred speeds in all tests.

The participant will mark the appropriate correct option on the computer screen with the help of the mouse, according to the warning coming from the headphones during walking.

Individuals' response accuracy will be used as an outcome measure.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Patients with Lung Cancer:

1. Individuals between the ages of 18-65
2. Individuals willing to participate in the research
3. Individuals diagnosed with lung cancer stage I-II-III
4. Individuals whose treatment has been completed and at least 6 months have passed since
5. Does not have any orthopedic problems that will prevent him from walking on the treadmill individuals
6. Having no problem in reading and/or understanding the scales and cooperating with the tests eligible individuals will be included in the study.

Inclusion Criteria for the Control Group:

1. Individuals between the ages of 18-65
2. Individuals willing to participate in the research
3. Individuals without a diagnosis of any lung disease
4. Does not have any orthopedic problems that will prevent him from walking on the treadmill individuals
5. Having no problem in reading and/or understanding the scales and being cooperative with the tests eligible individuals will be included in the study.

Exclusion Criteria:

Exclusion Criteria for Patients with Lung Cancer:

1. Individuals with the presence of metastases
2. Individuals with hearing problems
3. A neurological disease or other clinical diagnoses that may affect the cognitive status Individuals with disabilities will not be included in the study.

Exclusion Criteria for the Control Group:

1. Individuals with hearing problems
2. A neurological disease or other clinical diagnoses that may affect the cognitive status Individuals with disabilities will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients who were diagnosed with lung cancer at Liv Hospital Ankara were included in the study.
  Patients between the ages of 18-65 who are willing to participate will be taken. Snowball method will be used for the control group.
  Volunteer relatives of the patient and the researcher, and contact with hospital staff and then with other individuals in the same way.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Evaluating Dual Task Performance | 10 minutes
  Individuals' response accuracy will be used as an outcome measure.
Evaluation of Respiratory Muscle Endurance | 15 minutes
  It will be done with the Power Breathe device at 60% of the maximal inspiratory pressure at a fixed threshold load and the time the patient can sustain will be recorded. The resulting measurement is the product of the test time and the pressure measurement corresponding to the test time.

SECONDARY OUTCOMES:
Measurment of Tissue Oxygenation | 10 minutes
  Tissue oxygenation of the intercostal muscles during the respiratory muscle endurance test. The MOXY monitor will be used to measure tissue oxygenation of the intercostal muscles during the test. The Moxy monitor measures local oxygen saturation and total hemoglobin in muscle capillaries using the near infrared spectrum (NIRS).
Measurment of Fatigue | 5 minutes
  The fatigue severity scale, consisting of a total of 9 items, will be used. The individual should answer the questions by thinking about the last week. Each item is scored between 1 and 7. A total score of 36 and above or a scale score of 4 and above indicates severe fatigue in patients.
Measurment of Quality of Life | 5 minutes
  It will be evaluated by the European Organization for Cancer Research and Treatments (EORTC) QLQ-C30 questionnaire.
Physical Activity Level | 5 minutes
  It will be evaluated by International Physical Activity Questionnaire Short Form
Cognitive Function | 10 minutes
  It will be evaluated by The Montreal Cognitive Evaluation Scale. The highest score that can be obtained is 30 and the lowest score is 0. If the score is 21 or above, the individual's cognitive level is considered normal.

REFERENCES:
- [Result] Schabath MB, Cote ML. Cancer Progress and Priorities: Lung Cancer. Cancer Epidemiol Biomarkers Prev. 2019 Oct;28(10):1563-1579. doi: 10.1158/1055-9965.EPI-19-0221. PMID 31575553
- [Result] Ettinger DS, Akerley W, Borghaei H, Chang AC, Cheney RT, Chirieac LR, D'Amico TA, Demmy TL, Ganti AK, Govindan R, Grannis FW Jr, Horn L, Jahan TM, Jahanzeb M, Kessinger A, Komaki R, Kong FM, Kris MG, Krug LM, Lennes IT, Loo BW Jr, Martins R, O'Malley J, Osarogiagbon RU, Otterson GA, Patel JD, Pinder-Schenck MC, Pisters KM, Reckamp K, Riely GJ, Rohren E, Swanson SJ, Wood DE, Yang SC, Hughes M, Gregory KM; NCCN (National Comprehensive Cancer Network). Non-small cell lung cancer. J Natl Compr Canc Netw. 2012 Oct 1;10(10):1236-71. doi: 10.6004/jnccn.2012.0130. PMID 23054877
- [Result] Mustian KM, Sprod LK, Janelsins M, Peppone LJ, Mohile S. Exercise Recommendations for Cancer-Related Fatigue, Cognitive Impairment, Sleep problems, Depression, Pain, Anxiety, and Physical Dysfunction: A Review. Oncol Hematol Rev. 2012;8(2):81-88. doi: 10.17925/ohr.2012.08.2.81. PMID 23667857
- [Result] Anderson-Hanley C, Sherman ML, Riggs R, Agocha VB, Compas BE. Neuropsychological effects of treatments for adults with cancer: a meta-analysis and review of the literature. J Int Neuropsychol Soc. 2003 Nov;9(7):967-82. doi: 10.1017/S1355617703970019. PMID 14738279
- [Result] Falleti MG, Sanfilippo A, Maruff P, Weih L, Phillips KA. The nature and severity of cognitive impairment associated with adjuvant chemotherapy in women with breast cancer: a meta-analysis of the current literature. Brain Cogn. 2005 Oct;59(1):60-70. doi: 10.1016/j.bandc.2005.05.001. Epub 2005 Jun 21. PMID 15975700
- [Result] Boykoff N, Moieni M, Subramanian SK. Confronting chemobrain: an in-depth look at survivors' reports of impact on work, social networks, and health care response. J Cancer Surviv. 2009 Dec;3(4):223-32. doi: 10.1007/s11764-009-0098-x. Epub 2009 Sep 16. PMID 19760150
- [Result] Joly F, Giffard B, Rigal O, De Ruiter MB, Small BJ, Dubois M, LeFel J, Schagen SB, Ahles TA, Wefel JS, Vardy JL, Pancre V, Lange M, Castel H. Impact of Cancer and Its Treatments on Cognitive Function: Advances in Research From the Paris International Cognition and Cancer Task Force Symposium and Update Since 2012. J Pain Symptom Manage. 2015 Dec;50(6):830-41. doi: 10.1016/j.jpainsymman.2015.06.019. Epub 2015 Sep 5. PMID 26344551
- [Result] Lange M, Joly F, Vardy J, Ahles T, Dubois M, Tron L, Winocur G, De Ruiter MB, Castel H. Cancer-related cognitive impairment: an update on state of the art, detection, and management strategies in cancer survivors. Ann Oncol. 2019 Dec 1;30(12):1925-1940. doi: 10.1093/annonc/mdz410. PMID 31617564
- [Result] Hodgson KD, Hutchinson AD, Wilson CJ, Nettelbeck T. A meta-analysis of the effects of chemotherapy on cognition in patients with cancer. Cancer Treat Rev. 2013 May;39(3):297-304. doi: 10.1016/j.ctrv.2012.11.001. Epub 2012 Dec 6. PMID 23219452
- [Result] Falbo S, Condello G, Capranica L, Forte R, Pesce C. Effects of Physical-Cognitive Dual Task Training on Executive Function and Gait Performance in Older Adults: A Randomized Controlled Trial. Biomed Res Int. 2016;2016:5812092. doi: 10.1155/2016/5812092. Epub 2016 Dec 8. PMID 28053985
- [Result] Hofman M, Ryan JL, Figueroa-Moseley CD, Jean-Pierre P, Morrow GR. Cancer-related fatigue: the scale of the problem. Oncologist. 2007;12 Suppl 1:4-10. doi: 10.1634/theoncologist.12-S1-4. PMID 17573451
- [Result] Morrow GR. Cancer-related fatigue: causes, consequences, and management. Oncologist. 2007;12 Suppl 1:1-3. doi: 10.1634/theoncologist.12-S1-1. No abstract available. PMID 17573450
- [Result] Cankurtaran ES, Ozalp E, Soygur H, Ozer S, Akbiyik DI, Bottomley A. Understanding the reliability and validity of the EORTC QLQ-C30 in Turkish cancer patients. Eur J Cancer Care (Engl). 2008 Jan;17(1):98-104. doi: 10.1111/j.1365-2354.2007.00827.x. PMID 18181898
- [Result] Gencay-Can A, Can SS. Validation of the Turkish version of the fatigue severity scale in patients with fibromyalgia. Rheumatol Int. 2012 Jan;32(1):27-31. doi: 10.1007/s00296-010-1558-3. Epub 2010 Jul 24. PMID 20658235
- [Result] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Result] Anton HA, Miller WC, Townson AF. Measuring fatigue in persons with spinal cord injury. Arch Phys Med Rehabil. 2008 Mar;89(3):538-42. doi: 10.1016/j.apmr.2007.11.009. PMID 18295634
- [Result] Crum EM, O'Connor WJ, Van Loo L, Valckx M, Stannard SR. Validity and reliability of the Moxy oxygen monitor during incremental cycling exercise. Eur J Sport Sci. 2017 Sep;17(8):1037-1043. doi: 10.1080/17461391.2017.1330899. Epub 2017 May 30. PMID 28557670
- [Result] Tomporowski PD, Audiffren M. Dual-task performance in young and older adults: speed-accuracy tradeoffs in choice responding while treadmill walking. J Aging Phys Act. 2014 Oct;22(4):557-63. doi: 10.1123/japa.2012-0241. Epub 2013 Dec 4. PMID 24306656